CLINICAL TRIAL: NCT00793234
Title: Single Intravenous Administration of TB-402 for the Prophylaxis of Venous Thromboembolic Events (VTE) After Total Knee Replacement Surgery: A Dose-Escalating, Multicenter, Randomised, Active- Controlled Open Label Study
Brief Title: Single Intravenous Administration of TB-402 for the Prophylaxis of Venous Thromboembolic Events (VTE) After Total Knee Replacement Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ThromboGenics (Industry)
Collaborators: BioInvent International AB (Industry); Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TB-402-004
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Total Knee Replacement Surgery
Keywords: TKR; VTE; DVT
MeSH Terms: interventions — TB 402; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): 0.3 mg/kg TB-402
  Interventions: Drug: TB-402
- 2 (Experimental): 0.6 mg/kg TB-402
  Interventions: Drug: TB-402
- 3 (Experimental): 1.2 mg/kg TB-402
  Interventions: Drug: TB-402
- 4 (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: TB-402 — TB-402 administered as single bolus 18-24 post total knee replacement surgery.
  Arms: 1; 2; 3
Drug: Enoxaparin — Enoxaparin 40mg/day sc injection for at least 10 days post-surgery
  Arms: 4

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a single administration of TB-402 for the prevention of VTE in patients undergoing knee replacement surgery.

DETAILED DESCRIPTION:
Currently available anticoagulant therapies for the prevention of VTE include low molecular weight heparins, pentasaccharides and vitamin K antagonists, all of which have inherent limitations(1-3).

Improved anticoagulant agents are therefore required(4). A novel antithrombotic agent requires demonstration of both efficacy and safety in relevant populations. Phase II studies are frequently performed in patients undergoing total hip replacement and/or total knee replacement because of the high and well documented incidence of deep vein thrombosis in the absence of adequate thromboprophylaxis(5-7).

In this study, we assess the safety and efficacy of TB-402, a novel antithrombotic agent that partially inhibits factor VIII, in the prevention of VTE in patients undergoing total knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged > 18 and < 80 years old
* Female patients should be post menopausal
* Patients undergoing primary elective total knee replacement surgery
* Written informed consent obtained from the patient (or a legally acceptable representative) prior to inclusion in the study
* Willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* Body weight < 50 kg or > 100 kg
* Patients undergoing a hemiarthroplasty, surface repair or revisionary surgery of the knee
* Confirmed symptomatic deep vein thrombosis or pulmonary embolism within the past year
* Anticipated use of indwelling intrathecal or epidural catheter for more than 4 h after surgery or during the entire study
* Uncontrolled hypertension (SBP>160 mm Hg or DBP > 100 mm Hg)
* History of intracranial or intraocular bleeding. History of gastrointestinal and/or endoscopically verified ulcer disease within the past year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The occurrence of total bleeding defined as major and/or clinically relevant non-major bleeding events, from randomisation until the end of the study. | All visists from randomization to end of study
Composite of the occurrence of asymptomatic DVT as detected by bilateral venography and symptomatic VTE, i.e. DVT or fatal or non-fatal PE. | Prior to hospital discharge Day 7-11

SECONDARY OUTCOMES:
Incidence of major bleeding events | All visists from randomization to end of study
Incidence of clinically significant non-major bleeding events | All visits from randomization to end of study
Incidence of minor bleeding events | All visits from randomization to end of study
Incidence of all cause mortality | All visits from randomization to end of study
Incidence of adverse events | All visists from randomization to end of study

CONTACTS AND LOCATIONS:
Locations (35):
- Bulgaria (5):
  - SHAT of orthopedics, traumatology and surgery "Sv. Pantaleimon " - Pleven Department of Orthopaedics and Traumatology, Pleven
  - Dept. of Orthopedics, UMHAT "Saint George", Plovdiv
  - MHAT Rousse, Rousse
  - MHAT "Sveta Anna" AD - Sofia, Clinic of Orthopedics and Traumatology, Sofia
  - MHAT "Sv. Anna", Department of Orthopaedics and Traumatology, Varna
- Israel (8):
  - Asaf Harofeh MC, Beer-Yaakov
  - Soroka MC, Beersheba
  - Rambam MC, Haifa
  - Shaare Zedek MC, Jerusalem
  - Meir Medical Center (MC), Kfar Saba
  - Beilinson Hospital, Petah Tikva
  - Kaplan MC, Rehovot
  - Sourasky MC, Tel Aviv
- Latvia (3):
  - Ltd "Liepajas regionala slimnica", Liepāja
  - Ltd "Traumatologijas un ortopedijas slimnica", Riga
  - Vidzemes slimnica, Valmiera
- Poland (5):
  - Szpital Uniwersytecki im. dr. Antoniego Jurasza w Bydgoszczy Klinika Ortopedii i Traumatologii Narządu Ruchu, Bydgoszcz
  - Wojewódzki Szpital Specjalistyczny im. L. Rydygiera w Krakowie, Oddział Kliniczny Ortopedii i Traumatologii Narządu Ruchu, Krakow
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Klinika Ortopedii i Traumatologii, Podlaski
  - Samodzielny Publiczny Szpital Kliniczny nr 4 w Lublinie, Katedra i Klinika Ortopedii Traumatologii i Rehabilitacji, Trzemeszno Lubuskie
  - Wojewódzki Szpital Bródnowski Samodzielny Publiczny Zakład Opieki Zdrowotnej, Oddział Chirurgii Urazowo-Ortopedycznej i Rehabilitacji, Warsaw
- Romania (3):
  - Spitalul Clinic de Urgenta Sf. Ioan Bucuresti, Bucharest
  - Spitalul Clinic de Urgenta Prof. Dr. Octavian Fodor CLUJ NAPOCA, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Craiova, Craiova
- Russia (8):
  - Municipal Healthcare Institution "City Clinical Hospital No. 3", Chelyabinsk
  - Moscow State Healthcare Institution "City Clinical Hospital No. 15 n.a. O.M. Filatov", Moscow
  - Municipal Healthcare Institution "City Clinical Hospital No. 4", Orenburg
  - Saint Petersburg State Healthcare Institution "Aleksandrovskaya Hospital", Saint Petersburg
  - Federal State Medical Institution: Clinical Hospital #122 named after L.G. Sokolov under the Federal Medical-Biological Agency, Saint Petersburg
  - Saint Petersburg State Healthcare Institution "Municipal Multi-Speciality Hospital No. 2", Saint Petersburg
  - Federal State Institution "Russian Research Institute of Traumatology and Orthopedics n.a. R.R. Vreden under the Federal Authority for Healthcare and Social Development", Saint Petersburg
  - State Healthcare Institution "Samara Regional Clinical Hospital n.a. M.I. Kalinin", Samara
- Ukraine (3):
  - Cherkasska Regional Hospital. Department of Orthopedics and Traumatology., Cherkassy
  - Ivano-Frankіvsk Regional Clinical Hospital, Department of ortopedics and traumatology., Ivano-Frankivsk
  - Odessa Regional Clinical Hospital, Department of Orthopedics and Traumatology, Odesa